CLINICAL TRIAL: NCT04045886
Title: Conducting Perioperative Code Status and Goals of Care Discussions: A Bi-Institutional Study to Develop a Novel, Evidence-Based Curriculum for Anesthesiology Trainees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Richard D Urman, Associate Professor of Anesthesia, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2015P001375
Record Dates: First submitted 2017-11-13; First posted 2019-08-06 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Shared Decision Making; End of Life
MeSH Terms: conditions — Death | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Educational Modules group (Experimental): anesthesia residents are randomized to watch educational videos which is the intervention.
  Interventions: Behavioral: Online Educational Modules (Videos)
- Reading two research papers group (Active Comparator): anesthesia residents are randomized to read 2 research papers which is the active comparator
  Interventions: Behavioral: Online Educational Modules (Videos)

INTERVENTIONS:
Behavioral: Online Educational Modules (Videos) — 5 educational online modules (videos) about DNR/goals of care discussions that the participant will watch as part of the intervention. This is the only intervention.

SUMMARY:
Despite the importance of preoperative code status and goals of care discussion (CSD/GOCD), a formal curriculum for anesthesiology residents is lacking. Residents are often uncomfortable conducting these conversations and there is a lack of research investigating the effectiveness of formal, evidence-based teaching during anesthesia training. The investigators propose to develop a novel skills training program with the aims to assess its immediate effect on CSD/GOCD skills, long-term internalization of the CSD training, and the authenticity, feasibility and acceptability of the CSD program and observed standardized patient encounter (OSCE) interaction. In this prospective, randomized study, first year anesthesia residents will be assigned to the study or control group. Both groups will undergo pre- and post-intervention OSCEs. The control group will complete the online modules only, while the study group will complete the entire skills training program consisting of online modules, self-assessments, and small group exercises. To measure CSD/GOCD proficiency, all participants will interview trained patient actors in pre-and post intervention OSCE. Investigators will use existing scoring systems and surveys. Standard patient encounters will be video recorded and reviewed by two blinded clinician graders. The pre- and post-participation survey will assess comfort and experience with CSD/GOCD. The follow up surveys will assess long-term retention of training, comfort and interim experiences. Investigators will perform a validation of the existing CSD/GOCD assessment tools for use in the perioperative setting. If there is a clinically significant demonstrable benefit, investigators expect that the results will lead to a formalization of this innovative curriculum on a national scale.

DETAILED DESCRIPTION:
Despite the importance of code status discussions (CSD) and goals of care discussions (GOCD) before surgery, formal training for anesthesiology residents surrounding these patient interactions is lacking. Investigators propose to develop a novel CSD/GOCD skills training and testing program for anesthesiology residents. Resident participants will receive one of two educational interventions: a) online learning modules (Group A, Control group) or b) online learning modules followed by facilitated small group discussion and active learning exercises (Group B, Study group). All residents will undergo competency assessment of CSD and GOCD via an Objective Standardized Clinical Examination (OSCE). Accordingly, this study will test the central hypothesis that participants in the group with facilitated discussions and active learning will score more highly during the OSCE competency assessments immediately after training and at 3 and 6 months. Testing of this hypothesis will be accomplished through the following three Specific Aims:

1. Creation of a standardized CSD/GOCD Training Program:

   1. Online modules: This component of the training program will consist of online materials that can be consumed by residents at their convenience over the 3 week training period. Both Groups A and B will be given access to this material.
   2. Self-Assessment and Small group exercises: This component of the training program will consist of facilitated discussions, role playing, and guided reflective writing in order to advance upon the material received in the online training. Only Group B will receive this training prior to OSCE competency assessments.
2. Development and validation of a CSD/GOCD OSCE: Published best-practice principles for the development of OSCE competency assessments will be used to create separate experiences for CSD and GOCD. While keeping the core components of examinations the same, several clinical stems will be created for each OSCE to prevent recall bias.
3. Validation of the existing CSD/GOCD assessment tools for the perioperative setting: A previously described modified Delphi technique will be used to further develop the itemized and global assessment tools. Then, a standard setting method will be used to determine the minimum passing score (MPS) for the OSCE competency assessment.

EXPERIMENTAL DESIGN and METHODS:

Investigators will perform a prospective randomized controlled trial as detailed below. The overall hypothesis of this study is that anesthesiology residents who receive facilitated discussions and active learning will score more highly during the OSCE competency assessments immediately after training and at 3 and 6 months. This will be tested through the following Specific Aims:

1. Creation of a standardized CSD/GOCD Training Program: Investigators will develop a novel curriculum consisting of online modules covering the skills needed to Prepare for the Discussion, address Values and Goals of Care, explain Informed Consent for Code Status Discussions, and Summarize the Discussion for the patient. It will consist of evidence-based, best practices content covering professional (i.e. ASA) guidelines, current literature, and effective communication strategies. The Program will be completed over 1 week. Group A will receive the Online Modules components and Group B will receive two papers on CSD/GOCD topics.

   Online Modules: This component of the training program will consist of online materials that can be consumed by residents at their convenience over the 3 week training period. A series of short videos with lectures by various experts in the field which will include a detailed review of key scientific and educational research literature as well as a practical 'how-to' guide for CSD and GOCD.
2. Development and validation of a CSD OSCE and GOCD OSCE: Published best-practice principles for the development of OSCE competency assessments will be used to create separate experiences for CSD and GOCD. While keeping the core components of examinations the same, several clinical stems will be created for each OSCE to prevent recall bias.
3. Investigators will develop and validate a standardized OSCE curriculum with an input from a multidisciplinary team, including representatives from surgery, anesthesiology, palliative medicine, nursing, and chaplaincy. CSD/GOCD skills will be assessed using a validated Code Status Discussion Checklist. The training program will be based on previous work developing similar programs and simulation scenarios for the Operating Room Emergency Checklists. This program resulted in an increase from 75% of key items completed to 94%.
4. Case Development: Two case scenarios will be utilized, building on experience from our preliminary data. These were described in Preliminary Studies: both will be oncology patients with an active do not resuscitate (DNR) and no not intubate (DNI) order: One with cholecystitis presenting for a cholecystectomy, and the other with an impending pathological femur fracture presenting for an open reduction and internal fixation.
5. Validation and further development of existing CSD and GOCD assessment tools: A previously described modified Delphi technique will be used to create the itemized and global assessment tools. Then, a Standard Setting method will be used to determine the minimum passing score (MPS) for the OSCE competency assessment.

   a. Checklist Creation: i. Step 1: Engage a group of educational and content experts from at least 3 institutions to create the checklist items through a modified Delphi technique.

   ii. Step 2: Convene a face-to-face meeting of experts to perform an standard setting process to determine a minimum passing score (MPS).

   iii. Step 3: All OSCE performances will be videotaped and a group of raters will be engaged to grade all of the resident performances. Their ratings will be assessed for interrater and intra-rater reliability, which is one component of validity assessment.

   b. Training for Standardized Patients and Graders: Both the standardized patient and the graders will undergo training to familiarize them with the grading tools and the study scenarios.

   Assessment: Using validated tools, investigators will assess the impact of the study by analyzing the initial baseline survey, graded performance on Pre- and Post-Intervention OSCE, and the 3 and 6 month follow-up survey. Specific outcomes analyzed will include:
   * The immediate effect of the training program intervention on improving CSD/GOCD skills
   * Long-term effect and internalization of the CSD/GOCD training
   * The authenticity of the OSCE interaction
   * The feasibility and acceptability of the training program and OSCE

ELIGIBILITY:
Inclusion Criteria:

• Current Anesthesiology Resident at the Brigham and Women's Hospital

Exclusion Criteria:

* Not a current anesthesiology resident
* Prior study participation
* Unable to complete both OSCEs during a 1 week rotation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Performance on the assessment/scoring tool. | 1 week, includes evaluation during the OSCE examination, including both pre and post intervention OSCE
  Assessment tool was designed by the investigators for this study. The scoring tool measures conversation/communication skills based on 4 domains: general patient interviewing skills, discussing goals of care, discussing code status, and responding to emotion. The observed scale is 1-5 (low to high) for each domain. Scores will be then added for all domains to come up with a final score (possible range 4-20). Better values represent a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No